CLINICAL TRIAL: NCT00643422
Title: Reproducibility of Retinal Thickness and Volume Measurements Determined With the Cirrus Spectral Domain OCT
Brief Title: Reproducibility of Cirrus Optical Coherence Tomography Measurements
Status: Completed | Type: Observational
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Stefan Hagen, MD, Ludwig Boltzmann Institute of retinology and biomicroscopic laser surgery
Other Study IDs: Cirrus_OCT_0308
Record Dates: First submitted 2008-03-22; First posted 2008-03-26 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: normal eyes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observation
  Interventions: Device: Cirrus™ HD-OCT, Carl Zeiss Meditec AG

INTERVENTIONS:
Device: Cirrus™ HD-OCT, Carl Zeiss Meditec AG — the retinal thickness and volume is determined on two different days with the Cirrus™ HD-OCT.

SUMMARY:
In this study the reproducibility of optical coherence tomography measurements should be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* best corrected visual acuity of at least 20/25
* clear optical media

Exclusion Criteria:

* any kind of retinal pathology
* any kind of opacity of optical media
* any kind of intraocular surgery
* spherical refraction of more than 5 diopters
* cylindrical refraction of more than 3 diopters
* amblyopia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: attendants of health care center
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)

PRIMARY OUTCOMES:
retinal thickness | two

SECONDARY OUTCOMES:
retinal volume | two

CONTACTS AND LOCATIONS:
Locations (1):
- Rudolf Foundation Clinic, Vienna, Austria

REFERENCES:
- [Background] Wang XY, Huynh SC, Burlutsky G, Ip J, Stapleton F, Mitchell P. Reproducibility of and effect of magnification on optical coherence tomography measurements in children. Am J Ophthalmol. 2007 Mar;143(3):484-8. doi: 10.1016/j.ajo.2006.11.042. Epub 2006 Dec 22. PMID 17317392
- [Background] Paunescu LA, Schuman JS, Price LL, Stark PC, Beaton S, Ishikawa H, Wollstein G, Fujimoto JG. Reproducibility of nerve fiber thickness, macular thickness, and optic nerve head measurements using StratusOCT. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1716-24. doi: 10.1167/iovs.03-0514. PMID 15161831
- [Background] Polito A, Del Borrello M, Isola M, Zemella N, Bandello F. Repeatability and reproducibility of fast macular thickness mapping with stratus optical coherence tomography. Arch Ophthalmol. 2005 Oct;123(10):1330-7. doi: 10.1001/archopht.123.10.1330. PMID 16219723
- [Background] Danis RP, Fisher MR, Lambert E, Goulding A, Wu D, Lee LY. Results and repeatability of retinal thickness measurements from certification submissions. Arch Ophthalmol. 2008 Jan;126(1):45-50. doi: 10.1001/archopht.126.1.45. PMID 18195217
- [Background] Sadda SR, Tan O, Walsh AC, Schuman JS, Varma R, Huang D. Automated detection of clinically significant macular edema by grid scanning optical coherence tomography. Ophthalmology. 2006 Jul;113(7):1187.e1-12. doi: 10.1016/j.ophtha.2005.12.020. Epub 2006 May 2. PMID 16647123
- [Background] Budenz DL, Fredette MJ, Feuer WJ, Anderson DR. Reproducibility of peripapillary retinal nerve fiber thickness measurements with stratus OCT in glaucomatous eyes. Ophthalmology. 2008 Apr;115(4):661-666.e4. doi: 10.1016/j.ophtha.2007.05.035. Epub 2007 Aug 13. PMID 17706287
- [Background] Hsu SY, Tsai RK. Analysis of retinal nerve fiber layer and macular thickness measurements in healthy Taiwanese individuals using optical coherence tomography (Stratus OCT). J Glaucoma. 2008 Jan-Feb;17(1):30-5. doi: 10.1097/IJG.0b013e31811243b4. PMID 18303381
- [Background] Diabetic Retinopathy Clinical Research Network; Krzystolik MG, Strauber SF, Aiello LP, Beck RW, Berger BB, Bressler NM, Browning DJ, Chambers RB, Danis RP, Davis MD, Glassman AR, Gonzalez VH, Greenberg PB, Gross JG, Kim JE, Kollman C. Reproducibility of macular thickness and volume using Zeiss optical coherence tomography in patients with diabetic macular edema. Ophthalmology. 2007 Aug;114(8):1520-5. doi: 10.1016/j.ophtha.2006.10.055. Epub 2007 Mar 13. PMID 17353052
- [Derived] Hagen S, Krebs I, Haas P, Glittenberg C, Falkner-Radler CI, Graf A, Ansari-Shahrezaei S, Binder S. Reproducibility and comparison of retinal thickness and volume measurements in normal eyes determined with two different Cirrus OCT scanning protocols. Retina. 2011 Jan;31(1):41-7. doi: 10.1097/IAE.0b013e3181dde71e. PMID 20838360